CLINICAL TRIAL: NCT00695162
Title: Speech Intelligibility and Cognition: Are Inpatients Impaired by Noise?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Diana S. Pope, PhD, MS, RN, Principal investigator, Portland VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: #11-3307
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Auditory Perception; Memory; Hearing Impairment
Keywords: noise; speech intelligibility; cognition
MeSH Terms: conditions — Hearing Loss; Speech Intelligibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): hearing impaired inpatients
  Interventions: Other: quiet; Other: non-speech noise; Other: speech noise
- 2 (Other): Non-hearing-impaired inpatients
  Interventions: Other: quiet; Other: non-speech noise; Other: speech noise

INTERVENTIONS:
Other: quiet — no noise
Other: non-speech noise — noise without speech
Other: speech noise — noise with speech present

SUMMARY:
Study Objectives:

* 1. To examine the extent to which noise typical of nursing units reduces speech intelligibility in acutely ill hospitalized patients
* 2. To examine the extent to which noise typical of nursing units impairs recall in acutely ill hospitalized patients
* 3. To quantify severity of reduced performance associated with age, familiarity with the healthcare setting, hearing and health status.

Plan:

One hundred and twenty inpatients from the four medical/surgical nursing units at the Portland VA Medical Center, 60 with normal hearing and 60 with hearing impairment will be recruited to participate in the study. Following assessment to ascertain eligibility and obtaining informed consent, patients will be tested in a sound booth housed at the National Center for Rehabilitative Auditory Research (NCRAR). Designed so that each patient serves as his or her own control, we can accommodate considerable baseline variability between patients without adversely affecting required sample size. Patients' performance in speech intelligibility and recall tests will be measured using a constant level of speech, in controlled environments of no noise (baseline), white noise, hospital noise and hospital noise with speech, all delivered via headphones in pseudo-random order. Performance will be measured in each type of noise at decibel levels equivalent to those currently experienced on nursing units and at lower levels that prior studies have shown are more conducive to effective communication

By selecting measures that are particularly relevant to the safe care of hospitalized patients, and that have been studied extensively in healthy populations in highly controlled conditions, we expect to find compelling and unambiguous evidence that hospitalized patients correctly hear and recall very little of what is said to them during their hospitalizations. The majority of hospitalized patients stay on acute care nursing units during most or all of their hospitalizations, making this an appropriate population to study in the context of their responses to the noises typical in these environments. Perhaps most importantly, this study will heighten awareness of health-care personnel to the levels of impairment suffered by their patients - both in their ability to correctly interpret speech and to recall it - in the typical noisy environments of nursing units.

ELIGIBILITY:
Inclusion criteria:

* Adult inpatients on medical/surgical nursing units at the Portland VA, greater than 18 years of age will be eligible to participate.

Exclusion criteria for 60 participants with hearing impairment:

* Cognitively or physically unable to participate (reported by patient or nurse); electronic chart notes indicate patient exhibits aggressive behavior, documented dementia, Alzheimer's disease, or severe psychosocial disorder, patient undergoing detoxification, individual is not legally capable of independently providing informed consent
* Patients who are not native American English speakers.
* Patients who exhibit Meniere's disease or retrocochlear disorder based on patient report or notes in patient's chart.
* Patient exhibits active or recent history of middle ear disorder based on otoscopy, tympanometry, immittance or notes in patient chart; 5) patients unwilling to participate.

Exclusion criteria for the other 60 participants:

* Cognitively or physically unable to participate (reported by patient or nurse); electronic chart notes indicate patient exhibits aggressive behavior, documented dementia, Alzheimer's disease, or severe psychosocial disorder, patient undergoing detoxification, individual is not legally capable of independently providing informed consent
* Patients who are not native American English speakers.
* Patients who exhibit Meniere's disease or retrocochlear disorder based on patient report or notes in patient's chart.
* Patient exhibits active or recent history of middle ear disorder based on otoscopy, tympanometry, immittance or notes in patient chart.
* Patients with hearing loss that exceeds 25 dBHL in any frequency between .l5 and 3 kHz.
* Patients unwilling to participate.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in the percent of correctly identified words at different signal-to-noise rations (levels +4, +8 and +12 db) above that of the two types of noise, relative to the percent identified in quiet | immediately after presentation

SECONDARY OUTCOMES:
Change in the percent of correctly recalled words at different signal-to-noise rations (levels +4, +8 and +12 db) above that of the two types of noise, relative to the percent recalled in quiet | five minutes after presentation

CONTACTS AND LOCATIONS:
Overall Officials: Diana S Pope, PhD, MS, RN, Principal Investigator — Portland VA Medical Center
Locations (1):
- Portland VA Medical Center, Portland, Oregon, United States